CLINICAL TRIAL: NCT06467643
Title: Minimally Invasive Root Canal Treatment With Active Disinfection on Single Rooted Teeth With Periapical Lesions: A Preliminary Randomized Clinical Trial.
Brief Title: Minimally Invasive Root Canal Treatment With Active Disinfection on Single Rooted Teeth With Periapical Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint-Joseph University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: usj-2023-213
Record Dates: First submitted 2024-06-14; First posted 2024-06-21 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-06

CONDITIONS: Radiographic Healing of Periapical Lesions Following Ultrasonic Activation of Heated Sodium Hypochlorite Without Instrumentation of Root Canals
Keywords: Apical periodontitis; disinfection; healing; intracanal heating; minimally invasive endodontics; noninstrumentation; passive ultrasonic activation
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group IHAN (Experimental): The canal was irrigated with 5 mL room temperature 5.25% NaOCl and PUA was performed. Short vertical strokes were achieved for 30 seconds as manufacturer's instructions. After the first cycle of PUA, the canal was irrigated with 5 mL of 17% EDTA and kept in the canal for 60 seconds and then flushed out with 5 mL of saline. The root canal was filled again with 5.25% sodium hypochlorite and heated in the canal for 10 seconds using extra-fine heat carrier (0.04 taper) attached to a System B device. The temperature was fixed at 150 °C. Three consecutive cycles of PAU and intra-canal heating of sodium hypochlorite were performed. A final rinse of 5mL 17% EDTA was performed for 60 seconds followed by 5 mL of saline.
  Interventions: Procedure: non-instrumented root canal treatment with passive ultrasonic activation of heated sodium hypochlorite
- Group R-IHAN (Active Comparator): Each canal was prepared using Reciproc Blue nickel titanium primary file 25/08 (VDW, Munich, Germany) driven by a Xsmart IQ motor (Dentsply, Maillefer, Ballaigues, Switzerland) according to the manufacturer's instructions. Continuous checking of the canal patency was done using size 10 handfile followed by irrigation with 3 mL room temperature 5.25% sodium hypochlorite using irriflex endodontic irrigation needle mounted on a 3mL syringe each time the rotary file was removed out of the canal. Once the instrumentation was done, the canal was irrigated with 5 mL of 17% ethylenediaminetetraacetic acid (EDTA) kept for 60 seconds and then flushed with 5 mL of saline. NaOCl was placed in the canal and PUA followed by intracanal heating was performed three times as described for group 1 (IHAN).
  Interventions: Procedure: conventional root canal treatment with passive ultrasonic activation of heated sodium hypochlorite

INTERVENTIONS:
Procedure: non-instrumented root canal treatment with passive ultrasonic activation of heated sodium hypochlorite — Root canals were irrigated with room temperature 5.25% sodium hypochlorite which was activated ultrasonically for 30 seconds and then intra-canal heated using a heat carrier to a temperature fixed at 150 degree celsius. Three consecutive cycles of PAU and intra-canal heating of sodium hypochlorite were performed. After the first and the last cycle, root canals were irrigated with 5 mL of 17% ethylenediaminetetraacetic acid (EDTA) and kept in the canal for 60 seconds and then flushed out with 5 mL of saline. Root canals of this group were kept un-instrumented.
  Arms: Group IHAN
Procedure: conventional root canal treatment with passive ultrasonic activation of heated sodium hypochlorite — Root canals were convetionally prepared using Reciproc Blue rotary files according to the manufacturer's instructions. Once the instrumentation was done, the canal was irrigated with 5 mL of 17% ethylenediaminetetraacetic acid (EDTA) kept for 60 seconds and then flushed with 5 mL of saline. NaOCl was placed in the canal and PUA followed by intracanal heating was performed three times as described for group 1 (IHAN).
  Arms: Group R-IHAN

SUMMARY:
A novel form of root canal treatment RCT, referred as minimally invasive endodontics MIE, has emerged recently to adopt a unique approach that emphasize reducing tooth structural changes post-treatment (32). MIE seeks to maintain as much of the tooth's healthy coronal, cervical, and radicular anatomy as practical. Access opening, root canal cleaning and shaping, as well as surgical endodontics are all potential areas where MIE can be applied in endodontic therapy (34,36). Technological and technical progress, based on new tools, files and devices, are now allowing the simplification of this approach.

In the context of endodontics, the question may be whether conventional therapeutic approaches are minimally invasive enough (32,34), or whether a less invasive approach is required. This preliminary clinical study examined radiographically a minimally invasive shaping protocol combined with heated multi-sonic based irrigation to achieve disinfection with the removal of the least amount of dentin from the root's hard tissue during root canal shaping, compared to conventionally instrumented root canals, by focusing on the following aspects:

* The change in the area of the periapical lesion (measured in square millimeters) between T0, T3, T6 and T9
* The speed of repair of healed/healing periapical lesions (absolute speed of shrinkage and relative speed of shrinkage).

In addition, this study evaluated the association between radiographic outcomes and the type of endodontic treatment. Results obtained concerning the mentioned factors were compared across both techniques as well as the available ex-vivo and in vivo studies present in the literature. With the objective of cleaning and disinfecting the root canals as a complex while conserving root integrity, further efforts, to adopt such technique in posterior teeth where the mastication force and stress are at their most, could be done to set guidelines for an effective and more conservative root canal therapy.

DETAILED DESCRIPTION:
Microorganisms are the primary cause of pulp and periapical disorders (1). The key objective of endodontic therapy is to prevent or to heal apical periodontitis by eliminating inflamed and/or infected pulpal tissues and establishing aseptic intraradicular conditions conductive to periradicular healing (2). This goal is achieved by performing a chemo-mechanical debridement of the root canal system all while preserving the tooth's structural integrity for successful function (3,4).

Root canal instrumentation is primarily done to optimize irrigation and cleaning, particularly in the apical region, and to facilitate an hermetic obturation (5,6). However, mechanical instrumentation is linked with multiple drawbacks including the production of dentin debris and smear layer, the occurrence of iatrogenic errors, root structure weakening, and apical crack formation (7). It was also demonstrated that endodontic files are unable to touch the whole surface of the root canal walls due to the complexity of the root canal anatomy; affecting the total cleaning and the final prognosis (8). Accordingly, a variety of techniques and instruments can be used to render this step minimally invasive (9), as well as to improve the penetration of irrigants into the anatomical complexities (10,11). Minimally invasive endodontics MIE involves minimum intervention using smaller size and taper rotating files in combination with more effective irrigation protocols (12).

Ultrasonic activation of intracanal heated sodium hypochlorite NaOCl as a final irrigation protocol following root canal preparation showed superior bacterial reduction compared to canal preparation and NaOCl activation alone (13). Acoustic streaming and cavitation of heated irrigant are thought to be the working mechanisms (14,15). Recent in vitro studies have argued whether such irrigation protocols could be suitable to disinfect non-instrumented and/ or minimally tapered root canals (6,13,16).

Until now, no randomized clinical trials (RCTs) evaluated the in vivo efficacy of this protocol in un-instrumented canals. In the absence of sufficient models for clinical outcomes, only direct clinical studies evaluating both apical bone fill and tooth function/survival will offer compelling evidence regarding the efficacy of canal disinfection (4). Therefore, the aim of this preliminary randomized clinical trial was to evaluate radiographically the healing of periapical lesions on single rooted teeth following a non-instrumentation technique using ultrasonic activation with intracanal heating of sodium hypochlorite (IHAN) compared to rotary canal instrumentation and ultrasonic activation with heating of NaOCl (R-IHAN).

- Sample size: To determine the sample size, a power analysis for repeated-measures ANOVA (within-subjects factor with 4 measurements) was conducted using G*Power software 3.1.9.7 for Windows (Heinrich Heine, Universitat Düsseldorf, Düsseldorf, Germany); a power of 0.8, an alpha level of 0.05 were considered, and an effect size of 0.35 was calculated based on a previous study conducted by van der Borden et al (34). The minimum sample size required is 13 periapical lesions per group (26 in total). In order to account for losses to follow-up, an attrition rate of 20% was added, which results in a minimum total sample size of 32 (16 per group).

* Patient Selection Based on a power analysis for repeated-measures ANOVA (within-subjects factor with 4 measurements), the minimum sample size required is 13 periapical lesions per group (26 in total). In order to account for losses to follow-up, an attrition rate of 20% was added, which results in a minimum total sample size of 32 (16 per group). Patients with a noncontributory medical history were recruited at the Postgraduate Endodontics Clinic of the Faculty of Dentistry at the Saint Joseph University (Beirut-Lebanon) and were asked to sign a printed informed consent form after a detailed explanation of treatment procedures, possible outcomes, complications, and follow-up period desired. All selected teeth were single rooted maxillary and mandibular incisors, canines, or premolars with negative response on sensitivity testing and radiographic evidence of periapical bone loss of periapical index score PAI ≥3 according to the classification of Ørstavik et al. 1986. Only root canals in which stainless steel Kfile size 15 (Maillefer, Ballaigues, Switzerland) can passively reach the WL, an ultrasonic tip size 20/0.2 reaches the WL minus 3 to 4 mm, and the extra fine heat carrier tip (taper 4%) reaches the WL minus 4 to 5 mm, were included in this study. Pregnant women, teeth with broken or immature apices, resorption, calcifications, invading caries affecting the roots and abnormal mobility were excluded.
* Radiographic technique The included teeth were examined clinically and radiographically by using periapical radiography (PA) preoperatively (T0) and at recall (T3, T6 and T9). In order to take standardized radiographs throughout the experiment, pretreatment bite blocks were fabricated using a bite registration material (Kerr Corporation, Romulus, MI, USA) (Figure 1) and PA were taken standardized paralleling technique with number 2 periapical film (Durr Dental, Bietigheim-Bissingen, Germany) mounted on the customized radiographic stent and connected to the X-ray tube (Kodak RVG6100, Carestream Dental LLC, Atlanta, GA) via an adapter ring. The exposure parameters were 65 kV, 7.5 mA, and 0.15 seconds. Three experienced endodontists graded blindly and independently the pre-operative PAI of each sample according to the classification of Ørstavik et al. 1986. The lesion perimeter and area on the Xray were also measured in square and square millimeters respectively by using Image J 1.28 software (version 1.48v, National Institutes of Health, Washington, DC, USA) as previously described in multiple studies (7,18,19). Freehand selection was used to trace out the border of the lesion and then measure and record the area value. The examiners then met as a group to review all scores to enhance inter-rater agreement.
* Root canal procedure All treatments were performed in a single visit by a single endodontic postgraduate student. The full endodontic procedure was performed under strict aseptic setting and a dental operating microscope (Leica Microsystems, Wetzlar, Germany) at a x6.4 magnification. After confirming the clinical and radiological diagnosis, both the crown of the tooth as well as the clamp and the rubber dam were disinfected using hydrogen peroxide (6%), 5.25% sodium hypochlorite and 10% sodium thiosulfate respectively.

The access cavity was performed using sterile round diamond and endoZ burs (Maillefer, Ballaigues, Switzerland) mounted on a high-speed hand piece. An apex locator (Root ZX, J Morita Corp, Kyoto, Japan) and a size 15 stainless steel manual K-file (Maillefer, Ballaigues, Switzerland) were used to confirm the working length (WL) radiographically. The tooth was excluded from the study if the manual K-file size 15 was unable to reach WL passively.

The included teeth were randomly divided into 2 treatment groups by using random allocation software (http://www.randomization.com/) according to a standardized procedure: (1) Group IHAN (intracanal heating and passive ultrasonic activation of NaOCl only) (n=16): the canal was irrigated with 5 mL room temperature 5.25% NaOCl using irriflex endodontic irrigation needle (Produits Dentaires SA, Vevey, Switzerland) mounted on a 3mL syringe (Plastipak, Franklin Lakes, NJ, USA). PUA was performed using soft and flexible X silver tips (size 20/2%, length 21) mounted on an ultrasonic activator (Eighteeth, Changzhou Sifary Medical Technology Co., Ltd, Changzhou City, China) inserted in the canal to activate the solution. Short vertical up and down strokes were achieved for 30 seconds without breaching apical 2 mm as manufacturer's instructions. After the first cycle of PUA, an irriflex irrigation needle (Produits Dentaires SA, Vevey, Switzerland) mounted on a 3mL syringe (Plastipak, Franklin Lakes, NJ, USA) was used to irrigate the canal with 5 mL of 17% ethylenediaminetetraacetic acid (EDTA) and kept in the canal for 60 seconds and then flushed out with 5 mL of saline. The root canal was filled again with room temperature 5.25% sodium hypochlorite and heated in the canal for 10 seconds using extra-fine heat carrier (0.04 taper) attached to a System B device (Sybron dental, Orange, CA, USA) and moved with small in and out movements. The temperature was fixed at 150 °C. Both ultrasonic tip and heat carrier were introduced into the un-instrumented canal until binding then withdrawn 2-3 mm prior to activation and heating to avoid their wedging in the canal. Three consecutive cycles of PAU and intra-canal heating of sodium hypochlorite were performed. A final rinse of 5mL 17% EDTA was performed for 60 seconds followed by 5 mL of saline.

(2) Group R-IHAN (rotary instrumentation followed by intracanal heating and passive ultrasonic activation) (n=16): Each canal was prepared using Reciproc Blue nickel titanium primary file 25/08 (VDW, Munich, Germany) driven by a Xsmart IQ motor (Dentsply, Maillefer, Ballaigues, Switzerland) according to the manufacturer's instructions. Continuous checking of the canal patency was done using size 10 handfile followed by irrigation with 3 mL room temperature 5.25% sodium hypochlorite using irriflex endodontic irrigation needle mounted on a 3mL syringe each time the rotary file was removed out of the canal. Once the instrumentation was done, the canal was irrigated with 5 mL of 17% ethylenediaminetetraacetic acid (EDTA) kept for 60 seconds and then flushed with 5 mL of saline. NaOCl was placed in the canal and PUA followed by intracanal heating was performed three times as described for group 1 (IHAN).

After the completion of the endodontic procedures, gauging of the apex using K-flexofiles (Maillefer, Ballaigues, Switzerland) was done. each canal was dried with paper points and obturated with gutta-percha cones (Produits Dentaires SA, Vevey, Switzerland) and Kbiocer sealer (Rekita, Beirut, Lebanon). The largest well-adapted gutta-percha cone to the full WL without resistance was taken as master gutta-percha cone. A layer of 1 mm of glass ionomer (Fuji II LC Capsules, GC America, Alsip, IL, USA) was placed over the gutta percha in the pulp chamber and covered by layer of temporary filling material. A final periapical Xray was taken.

- Evaluation Recall checkup appointments were regularly scheduled every 3-6- and 9 months (20-22). Much care was taken to reach a high recall rate. Two patients out of 32 did not show on all the recall checkup appointments, hence they were excluded from the study (N=30), making the n=16 for IHAN and n=14 for R-IHAN. At recall examination, pain, swelling, sinus tract, gingival palpation, tenderness to percussion, and the quality of coronal restorations were recorded. Post-operative standardized radiographs were taken in order to monitor the healing of the periapical lesion. The lesion perimeter and area at the first visit were compared with those at recall, and each sample was given a post-operation PAI at T9.

Based on the area percentage change of lesions, the treatment outcome was presented in four categories: undetected lesion, reduction, enlargement, or unchanged. Reduction and enlargement of the radiolucency were determined only when the change in size of radiolucency was 20% or more (41)(42). An unchanged lesion was defined as a lesion change less than 20% (18). Treatment outcome scores with PAI were adjusted to reflect clinical success (PAI1 and PAI2 at follow-up), uncertain (PAI3 at follow-up for initial PAI4,5) and failure (persisting PAI3 and any PAI4 or PAI5 at follow-up). Failure was also recorded if the patient did not appear at any follow up recalls, a tooth had been extracted, or had evidence of a sinus tract involving the periapical area at recall (23). In order to assess the speed of repair of healed/healing periapical lesions (24), two formulas were used: (1) Absolute speed of shrinkage (mm2/day) = (initial detected area - final area) / duration of treatment; (2) Relative speed of shrinkage (/day) = (initial detected area - final area) x 100 / initial detected area x duration of treatment.

Statistical analysis The IBM SPSS Statistics software version 25.0 was used for data analysis. A P-value of less than 0.05 was considered statistically significant (P<0.05). Descriptive statistics were conducted; quantitative variables are presented as means and standard deviations, while qualitative variables are expressed as frequencies and percentages. One-sample T-tests and Wilcoxon signed-rank tests were employed to compare the percentage change in perimeter, surface, and opacity with a 20.0% threshold at T3. Student's T-tests and Mann-Whitney tests were utilized to identify significant differences in perimeter percentage change and surface percentage change between the techniques at T3, T6, and T9. A Friedman two-way test was employed to assess significant differences in perimeter and surface percentage change over time for the different techniques. The Mann-Whitney test was also employed to assess differences in absolute and relative speed between the different techniques. Chi-square (or Fisher's exact test) was utilized to analyze the relationship between the technique and final observed changes in terms of perimeters, surface, as well as treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy patients aging from 18 to 40 years old without any known allergic reactions or systemic diseases.
2. Mature necrotic single rooted teeth with a single canal.
3. Fully formed intact root apices.
4. Root canals in which stainless steel Kfile size 15 (Maillefer, Ballaigues, Switzerland) can passively reach the WL.
5. Root canals in which the chosen ultrasonic tip size 20/0.2 reaches the WL minus 3 to 4 mm (Figure 3) and the extra fine heat carrier tip (taper 4%) reaches the WL minus 4 to 5 mm.
6. Estimated working length 20-23 mm
7. Absence of canal calcifications.
8. Absence of root fracture and/or resorption.
9. Teeth with pre-operative periapical radiolucency and PAI score ≥3 according to the classification of Ørstavik et al. 1986.

Exclusion Criteria:

1. Roots with broken or immature open apices.
2. Roots presenting internal, external, or apical resorption.
3. Teeth with previous root canal treatment
4. Teeth with retracted or calcified canals.
5. Teeth with two canals or any other anatomic variations.
6. Extensively restored and prepared teeth.
7. Teeth invaded by caries affecting the roots.
8. Root length less than 16 mm.
9. Abnormal mobility of the tooth.
10. Patients with chronic generalized periodontitis
11. Pregnant patients
12. Patients younger than 18 years old

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2023-07-07 (Actual); Primary Completion 2023-10-07 (Actual); Study Completion 2024-04-07 (Actual)

PRIMARY OUTCOMES:
radiographic healing based of the area percentage change of lesions | 9 months
  the treatment outcome was presented in four categories: undetected lesion, reduction, enlargement, or unchanged. Reduction and enlargement of the radiolucency were determined only when the change in size of radiolucency was 20% or more. An unchanged lesion was defined as a lesion change less than 20%.
radiographic healing based on the periapical index score by Ørstavik et al. 1986 | 9 months
  Treatment outcome scores with PAI were adjusted to reflect clinical success (PAI1 and PAI2 at follow-up), uncertain (PAI3 at follow-up for initial PAI4,5) and failure (persisting PAI3 and any PAI4 or PAI5 at follow-up). Failure was also recorded if the patient did not appear at any follow up recalls, a tooth had been extracted, or had evidence of a sinus tract involving the periapical area at recall.

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Joseph University, Beirut, Lebanon